CLINICAL TRIAL: NCT03904303
Title: Test of a New Gel-based Colon Cleansing Agent Compared to Moviprep. A Randomized Single-blinded Cross-over Study
Brief Title: Test of a New Gel-based Colon Cleansing Agent Compared to Moviprep
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: REG-014-2018
Record Dates: First submitted 2019-01-29; First posted 2019-04-05 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Pharmacological Action

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geloprep (Experimental): Novel and patented Polyethylene glycol 3350 mixture
  Interventions: Drug: A 06 ad
- Moviprep (Active Comparator): Standard of care Polyethylene glycol 3350 mixture
  Interventions: Drug: A 06 ad

INTERVENTIONS:
Drug: A 06 ad — Colonic cleansing before colonoscopy and CT colonografi

SUMMARY:
Crossover study comparing Moviprep (for bowel cleansing) with a new gel-based colon cleansing agent before colonoscopy

DETAILED DESCRIPTION:
Crossover study comparing Moviprep (for bowel cleansing) with a new gel-based colon cleansing agent before colonoscopy.

Study performed in health subjects.

ELIGIBILITY:
Inclusion Criteria:

- Healthy

Exclusion Criteria:

* Allergy to content of products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel preparation scale (BBPscale) | Performed during the endoscopy procedure
  Visual assessment of the degree of bowel cleansing performed by the endoscopist (blinded). Right colon, colon transversum, and left colon are each judged on a scale from 0-3 with higher scores indicating better cleansing. Range of score between 0-9.
Adverse events related to intervention | Assessed 4 hours after last intake of cleansing product
  Any adverse event related to the intervention observed by investigators or as reported by the participant

SECONDARY OUTCOMES:
Blood pressure | Measured immediately before the colonoscopy starts, and every 5 minutes during colonoscopy and immediately after the end of the examination
  mmHg systolic and diastolic measured on right or left arm.
Saturation | Measured immediately before the colonoscopy starts, and every 5 minutes during colonoscopy and immediately after the end of the examination
  Oxymeter measuring the saturation of hemoglobin with oxygen as a percentage of 0-100%.
Heart rate | Measured immediately before the colonoscopy starts, and every 5 minutes during colonoscopy and immediately after the end of the examination
  Heart rate
Respiration frequency | Measured immediately before the colonoscopy starts, and every 5 minutes during colonoscopy and immediately after the end of the examination
  Respiration frequency

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, Professor MD, Study Chair — Department of Surgery, Zealand University Hospital
Locations (1):
- Zuh, Køge, Region of Zealand, Denmark